CLINICAL TRIAL: NCT04622943
Title: ShootSafe: An Interactive Web Platform to Teach Children Hunting, Shooting and Firearms Safety
Brief Title: An Interactive Web Platform to Teach Children Hunting, Shooting and Firearms Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, David Schwebel, University Professor of Psychology & Associate Vice President for Research Facilities & Infrastructure, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01CE003307 (NIH)
Record Dates: First submitted 2020-10-26; First posted 2020-11-10 (Actual); Results first posted 2025-03-10 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Safety Issues; Injuries; Firearm Injury
MeSH Terms: conditions — Wounds and Injuries | interventions — Nutritional Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- firearms safety (Experimental): Children will spend two 45-minute sessions engaged on ShootSafe, an internet-based training program on firearms safety.
  Interventions: Behavioral: firearms safety
- nutrition (Active Comparator): Children will spend two 45-minute sessions engaged in vHappy, an internet-based training program on nutrition and wellbeing.
  Interventions: Behavioral: nutrition

INTERVENTIONS:
Behavioral: firearms safety — interactive and engaging website with videos and educational games to teach children firearms, hunting and shooting safety
  Arms: firearms safety
Behavioral: nutrition — interactive and engaging website with videos and educational games to teach children about nutrition and wellbeing
  Arms: nutrition

SUMMARY:
Firearms injuries present a major pediatric public health challenge, killing >800 children ages 0-15 annually and leading to lifelong disability among >1000 survivors. About ⅓ of firearms injuries to children under age 15 are due to unintentional causes rather than suicide or homicide. The investigators propose development and evaluation of ShootSafe, an innovative, engaging, and educational website accessible by smartphone, tablet or computer that engages children to learn firearms safety.

ShootSafe extends existing programs to achieve 3 primary goals: a) teach children knowledge and skills they need to hunt, shoot, and use firearms safely; b) help children learn and hone critical cognitive skills of impulse control and hypothetical thinking needed to use firearms safely; and c) alter children's perceptions about their own vulnerability and susceptibility to firearms-related injuries, the severity of those injuries, and their perceived norms about peer behavior surrounding firearms use. ShootSafe will accomplish these goals through a combination of interactive games plus podcast videos delivered by peer actors (impactful testimonials about firearms injuries/deaths they experienced) and experts (wisdom & experience from trusted role models). The website will also incorporate brief messaging to parents, who will absorb key lessons and reinforce them with their children.

The website will be evaluated through a randomized controlled trial with 162 children ages 10-12, randomly assigning children to engage in the ShootSafe website or an active control website on child nutrition. The investigators will incorporate sub-aims to evaluate changes in children's (a) knowledge, (b) cognitive skills in impulse control and hypothetical thinking, (c) perceptions about firearms safety, and (d) simulated behavior when handling, storing and transporting firearms. All outcome measures will be assessed at baseline, immediately post-intervention, and at a 4-month follow-up assessment to evaluate retention. Training will comprise two 30-minute sessions.

ELIGIBILITY:
Inclusion Criteria:

* children ages 10-12 years
* English-speaking child and parent
* Experience or exposure to firearms in their homes or through engagement in hunting or shooting

Exclusion Criteria:

* disabilities that prohibit participants from valid understanding of or participation in the experimental protocol
* siblings of enrolled child

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 163 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Schwebel, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Youth Safety Lab, University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with qualified parties upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: after all primary analyses are conducted and published, for 3 year period
Access Criteria: qualified user with appropriate training and approval

REFERENCES:
- [Derived] Schwebel DC, Long DL, Johnston A, He Y, Morgan CH, Severson J, Taylor G, Trullinger K. Evaluation of ShootSafe, an Interactive, Sequential Website to Teach Youths Firearms Safety: A Randomized Clinical Trial. Am J Public Health. 2025 Dec;115(12):1971-1977. doi: 10.2105/AJPH.2025.308267. Epub 2025 Sep 18. PMID 40966575
- [Derived] Schwebel DC, Long DL, Gowey M, Severson J, He Y, Trullinger K. Study protocol: developing and evaluating an interactive web platform to teach children hunting, shooting and firearms safety: a randomized controlled trial. BMC Public Health. 2021 Feb 6;21(1):308. doi: 10.1186/s12889-021-10345-3. PMID 33549072

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Firearms Safety | Nutrition
Started | 83 | 80
Post-intervention Assessment | 77 | 75
Completed | 72 | 72
Not Completed | 11 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Firearms Safety | Nutrition | Total
Number analyzed (Participants) | 83 | 80 | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.4 (0.88) | 11.4 (0.78) | 11.4 (0.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 34 | 63
  Male | 54 | 46 | 100
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White/Caucasian | 57 | 54 | 111
  Race: African-American/Black | 24 | 22 | 46
  Race: Asian-American | 0 | 2 | 2
  Race: Native American/American Indian/Alaskan Native | 1 | 0 | 1
  Race: Chose not to report or missing | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latinx | 1 | 0 | 1
  Ethnicity: not Hispanic or Latinx | 80 | 77 | 157
  Ethnicity: Chose not to report or missing | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 83 | 80 | 163

OUTCOME MEASURES:

1. Primary Outcome: Number of Knowledge Items Answered Correctly
Description: firearms safety knowledge scale (10 items, minimum value 0 and maximum value 10). Higher scores indicate greater knowledge.
Time Frame: 1 week after intervention completed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Firearms Safety | Nutrition
Number analyzed (Participants) | 77 | 75
score on a scale | 8.2 (0.2) | 6.2 (0.2)

2. Primary Outcome: Risky Behavior in Simulated Hunting Scenario
Description: Number of simulated situations when it was dangerous to shoot the toy firearm and the child took shots
Time Frame: 1 week after intervention completed
Measure: Mean (Standard Deviation); unit: scenarios
Arm/Group | Firearms Safety | Nutrition
Number analyzed (Participants) | 77 | 75
scenarios | 1.8 (0.2) | 2.9 (0.2)

ADVERSE EVENTS:
Time Frame: 4 months
Description: Definitions do not differ from clinicaltrials.gov definitions.
Arm/Group | Firearms Safety | Nutrition
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/80
Other Adverse Events (participants affected / at risk) | 0/83 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-11): https://cdn.clinicaltrials.gov/large-docs/43/NCT04622943/Prot_SAP_000.pdf